CLINICAL TRIAL: NCT02186028
Title: Effect Of Oral Daily Supplementation With 400 IU Vs 200 IU Of Vitamin D In Term Healthy Newborns: A Randomised Control Trial
Brief Title: Effect of Oral Daily Supplementation With 400 IU Vs 200 IU of Vitamin D in Term Healthy Neonates
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lady Hardinge Medical College (Other Government)
Responsible Party: Principal Investigator, Sushma Nangia, M.D., Dr Sushma Nangia, M.D., D.M. (neonatology), Lady Hardinge Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LHMC/094/2012/VitD
Record Dates: First submitted 2014-07-07; First posted 2014-07-10 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Vitamin D Deficiency
Keywords: oral daily supplementation with vitamin D for 6 months
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D 400 IU (Experimental): Vitamin D-400IU/ml- 1ml daily
  Neonates will be administered Vitamin D 400 IU orally daily by the mother or other caregiver for a period of six months. The neonates will be followed up for compliance at 2 weeks, 6, 10 and 14 weeks and thereafter at 6 months of age.
  Interventions: Drug: Vitamin D
- Vitamin D 200IU (Active Comparator): Vitamin D 400IU/ml : 0.5ml daily
  Neonates will be administered Vitamin D 200 IU orally daily by the mother or other caregiver for a period of six months. The neonates will be followed up for compliance at 2 weeks, 6, 10 and 14 weeks and thereafter at 6 months of age.
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — Vit D 400 IU vs. Vit D 200 IU

SUMMARY:
The purpose of the study is to evaluate the effect of daily oral supplementation with vitamin D on serum Vitamin D levels in term healthy newborns. It has been found in various studies that vitamin D is highly deficient in Indian mother infant diads. There is a need to supplement vitamin D from neonatal period to prevent various metabolic disturbances due to vitamin D deficiency in later life. This study aims to find the effectiveness and the optimum dose of routine vitamin D supplementation in healthy term newborns for fulfilling the normal requirements in Indian infants.

DETAILED DESCRIPTION:
Vitamin D deficiency is highly prevalent in India as reported in various studies. Vitamin D supplementation is necessary as vitamin D is required not only for prevention of rickets as traditionally thought, but also for its emerging role in development of diseases such as myopathic disorders, proneness to infection, autoimmune disorders and cancers .However supplementation studies are limited and predominantly from foreign countries. Moreover most of them report variable outcomes with no unanimous outcome with respect to optimum dose and duration of supplementation of vitamin D. Various national authorities recommend different doses of vitamin D for supplementation. American Academy of Pediatrics, The Institute of Medicine of National Academics, The Drug and Therapeutics Committee of the Lawson Wilkins Pediatric Endocrine Society, the Canadian Pediatric Society and European Society for Pediatric Endocrinology recommend that 400IU of vitamin D should be supplemented in all infants starting from within a few days of birth throughout childhood. ESPGHAN recommends 800-1000 IU for high risk infants, Ireland recommends 200IU vitamin D per day, UK does not recommend any supplements upto 6 months of age , however if formula milk intake <500ml/day then 300 IU is recommended. There are no such guidelines for India. Hence this study aims at evaluating the proportion of vitamin D deficient

ELIGIBILITY:
Inclusion Criteria:

* Gestation > 37 weeks
* Birth weight >2.5 kg
* Informed consent of one of the parents
* Place of residence<10km

Exclusion Criteria:

* Presence of gross congenital malformation
* Need of resuscitation at birth
* Need for admission to neonatal ICU
* Refusal of consent

Ages: 2 Hours to 48 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2014-07; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Difference in vitamin D levels attained after oral supplementation with 400IU/day Vs 200IU/day of vitamin D for 6 months | 6 months

SECONDARY OUTCOMES:
Proportion of vitamin D deficient term healthy neonates at birth | at birth
  serum vitaminD levels > 20 ng/ml - sufficient 15 - 20 ng/ml - insufficient <15 ng/ml - deficient

OTHER OUTCOMES:
Proportion of neonates having vitamin D sufficiency after supplementation | 6 months
  serum vitamin D levels > 20 ng/ml - sufficient 15 - 20 ng/ml - insufficient <15 ng/ml - deficient
Proportion of neonates having vitamin D deficiency after supplementation | 6 months
  serum vitamin D levels > 20 ng/ml - sufficient 15 - 20 ng/ml - insufficient <15 ng/ml - deficient

CONTACTS AND LOCATIONS:
Overall Officials: Sushma Nangia, MD, DM, Study Chair — Lady Hardinge Medical College & Kalawati Saran Children's Hospital; Arvind Saili, MD, Study Director — Lady Hardinge Medical College & Kalawati Saran Children's Hospital
Locations (1):
- Kalawati Saran children's Hospital, Lady Hardinge Medical College, New Delhi, New Delhi, India